CLINICAL TRIAL: NCT00598377
Title: Assessment of Adrenal Functions in Patients With Autosomal Dominant Polycystic Kidney Disease
Brief Title: Adrenal Functions in Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Tevfik Ecder, Istanbul University, Istanbul Medical Faculty, Division of Nephrology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007/233; 2007/233
Record Dates: First submitted 2007-12-31; First posted 2008-01-21 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2008-02

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Autosomal dominant polycystic kidney disease; Adrenal functions; Renal volume; Glomerular filtration rate; Adrenal Cortex Function Tests
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Cosyntropin; adrenocorticotropin zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients with autosomal dominant polycystic kidney disease
  Interventions: Drug: Tetracosactin
- 2 (Active Comparator): Healthy subjects
  Interventions: Drug: Tetracosactin

INTERVENTIONS:
Drug: Tetracosactin — 1 microgram tetracosactin, intravenous injection, once for the test
  Other Names: Synacthen

SUMMARY:
We aimed to evaluate the hypothalamus-pituitary-adrenal axis in autosomal dominant polycystic kidney disease (ADPKD) patients. Twenty two ADPKD patients and 27 healthy subjects were enrolled.

DETAILED DESCRIPTION:
CONTEXT: Autosomal dominant polycystic kidney disease (ADPKD) is the most common hereditary kidney disease and extrarenal manifestations may be observed in many organ systems. Hypothalamus-pituitary-adrenal axis in patients with ADPKD was not evaluated extensively.

OBJECTIVE: We aimed to evaluate the hypothalamus-pituitary-adrenal axis in ADPKD patients.

METHODS: Twenty two ADPKD patients and 27 healthy subjects were enrolled. Basal dehydroepiandrosterone-sulfate (DHEAS) levels and cortisol and dehydroepiandrosterone responses to low dose short adrenocorticotropin stimulation test were assessed. Correlation analyses of these parameters with glomerular filtration rates, renal volumes and pain characteristics in patients with ADPKD were done.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Diagnosis of autosomal dominant polycystic kidney disease

Exclusion Criteria:

* A glomerular filtration rate below 60 ml/min
* History of recent major surgery
* Systemic infections with fever
* Significant hirsutism (Ferriman Gallwey score≥8)
* Congenital adrenal hyperplasia
* Late onset congenital adrenal hyperplasia
* Systemic corticosteroid use (including previous use)
* Topical corticosteroid use
* Menstrual irregularity
* History of thromboembolism
* Uncontrolled diabetes or hypertension
* History of psychosis
* Pregnancy
* Lactation
* History of hypersensitivity to tetracosactin

Ages: 20 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Inadequate response to tetracosactin infusion | 30 and 60 minutes after the drug is administered

CONTACTS AND LOCATIONS:
Overall Officials: Tevfik Ecder, Professor, Principal Investigator — Istanbul University, Istanbul Medical Faculty, Department of Internal Medicine, Division of Nephrology; Fatih Tufan, Fellow, Study Director — Istanbul University Istanbul Medical Faculty Department of Internal Medicine; Neşe Çolak, Professor, Study Director — Istanbul University Istanbul Medical Faculty Department of Internal Medicine Division of Endocrinology; Bora Uslu, Fellow, Study Chair — Istanbul University Istanbul Medical Faculty Department of Internal Medicine; Kültigin Türkmen, Fellow, Study Chair — Istanbul University Istanbul Medical Faculty Department of Internal Medicine; Mükremin Uysal, Fellow, Study Chair — Istanbul University Istanbul Medical Faculty Department of Internal Medicine; Nilüfer Alpay, Fellow, Study Chair — Istanbul University Istanbul Medical Faculty Department of Internal Medicine; Rian Dişçi, Professor, Study Director — Istanbul University Istanbul Medical Faculty Department of Public Health; Bledi Çerkezi, Fellow, Study Chair — Istanbul University Istanbul Medical Faculty Department of Radiology
Locations (1):
- Istanbul Univetsity, Istanbul Medical Faculty, Department of Internal Medicine, Istanbul, Turkey (Türkiye)